CLINICAL TRIAL: NCT05564871
Title: The Effectiveness of Occupational Therapy Teleintervention for Children Aged 5-8 With Neurodevelopmental Disorders.
Brief Title: Effectiveness of Occupational Therapy Teleintervention in Pediatric
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Stav Ben Zagmi, Occupational therapist, Hebrew University of Jerusalem
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HebrewHJ
Record Dates: First submitted 2022-09-14; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Telerehabilitation; Neurodevelopmental Disorders
Keywords: Telemedicine, NDD's, Occupational Therapy
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupation-based teleintervention (Experimental): 20 children and their parents will be participate in Occupation-based teleintervention.
  Interventions: Other: occupation-based teleintervention
- Occupation-based in person intervention (Experimental): 20 children and their parents will be participate in Occupation-based in person intervention.
  Interventions: Other: occupation-based teleintervention

INTERVENTIONS:
Other: occupation-based teleintervention — Intervention protocol will include 12 weekly based on the principles of the CO-OP approach. The intervention will focus on solving problems in the participant's daily life and implementing strategies in accordance with the goals set according to the COPM (Law et al., 2017). In the research group, the intervention will be carried out through videoconference sessions between an occupational therapist located at one of the child development units and the participant and their parents who are at home. The control group will receive a weekly session of CO-OP intervention in-person in one of the child development units.

SUMMARY:
The high prevalence of children with neurodevelopmental disorders (NDD's; 5-29%) combined with the low accessibility and availability of child development services in Israel raises an urgent need to develop innovative, effective and accessible models of intervention. Teleintervention is an innovative and practical option for providing developmental services, however the evidence for its effectiveness among this population are insufficient. Study goals are: (1) to adapt an occupation therapy intervention for remote delivery; (2) to assess its feasibility (in terms of adherence, treatment fidelity and satisfaction with care); (3) to assess its efficacy in promoting personal functional goals, participation in daily activities and QOL in children aged 5-8 years with NDD's. We will conduct a controlled study without randomization using mixed methods. Participants will include 40 children with NDD's and functional difficulties in daily life that will assigned to study group (teleintervention; n=20) or control group (in person intervention; n=20). The intervention program will include 12 weekly sessions based on an evidence-based approach (CO-OP), that will take place in videoconference or in personal meetings formats. The main outcome measures will include standard assessment tools aim to assess participation and QOL. Feasibility will be assessed in terms of adherence, fidelity and satisfaction with care using a descriptive statistics and feedback interviews. Effectiveness will be evaluated by group X time interaction using a repeated measure MANOVA. To examine the variables that predict adherence and success in treatment, linear regression will be used. In addition, a thematic analysis of the qualitative information will be performed.

DETAILED DESCRIPTION:
Background and aims: The high prevalence of children with neurodevelopmental disorders (NDD's; 5-29%) combined with the low accessibility and availability of child development services in the south region of Israel raises an urgent need to develop innovative, effective and accessible models of intervention. Teleintervention is an innovative and practical option for providing developmental services for people who are in their home, however the evidence for its effectiveness among this population are insufficient. Study goals are: (1) to adapt an occupation therapy intervention for remote delivery; (2) to assess its feasibility (in terms of adherence, treatment fidelity and satisfaction with care); (3) to assess its efficacy in promoting personal functional goals, participation in daily activities and QOL in children aged 5-8 years with NDD's. Methods: We will conduct a controlled study without randomization using mixed methods. Participants will include 40 children with NDD's and functional difficulties in daily life that will assigned to study group (teleintervention; n=20) or control group (in person intervention; n=20). Participants will be recruited from the child development unites at "Meuhedet" HMO in the southern district. The intervention program will include 12 weekly sessions based on an evidence-based approach (CO-OP), that will take place in videoconference or in personal meetings formats. The purpose of the intervention model is to improve personal goals that will be defined by each child and his/her parents. The main outcome measures will include standard assessment tools aim to assess participation and QOL. Participants will undergo baseline and post-intervention assessments. Feasibility will be assessed in terms of adherence, fidelity and satisfaction with care using a descriptive statistics and feedback interviews. Effectiveness will be evaluated by group X time interaction using a repeated measure MANOVA. To examine the variables that predict adherence and success in treatment, linear regression will be used. In addition, a thematic analysis of the qualitative information will be performed. Preliminary results from a pilot study (N= 14) conducted during the COVID-19 pandemic and military escalation demonstrated the feasibility of occupation therapy teleintervention. The results also suggest the protentional efficacy of the program, thus a clinically significant improvement was achieved in 80% / 73.68% of the personal goals practiced during the treatment according to the child and parent report (respectively). Expected results: the results of the study could constitute a theoretical and practical infrastructure for the establishment of occupational therapy teleintervention services in addition to face-to-face services that currently exist exclusively, for the large population of children with NDD's and to allow immediate implementation of the intervention program as part of the child development services in Israel. Importance to Medicine: This innovative, cost-effective format will improve accessibility to occupational therapy services for children with NDD's and their families in the peripheral regions of Israel. In the long run, it can be assumed that the integration of accessible and effective services in child development units will help reduce the burden on their families, promote their functioning and reduce the need for medical and social assistance services in the future.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew at mother tongue level
* Child's ability to identify at least three functional difficulties for the purpose of setting treatment goals
* Availability of computer with web camera and an IPad connected to broadband or Wi-Fi in their home

Exclusion Criteria:

* Children with somatic or physical disabilities, children diagnosed with ASD, following a brain injury or children with mental health disorders.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure - COPM (Law et al., 2017) | Change from baseline occupational performance at 6 months
  Hebrew version. The COPM is a widely used valid outcome measure in rehabilitation research, designed to measure the clients' self-perceptions of their activity performance and satisfaction with performance and detect changes over time. Participants in collaboration with the parents will be asked to identify goals and then rate their performance and satisfaction with performance on a scale of 1 to 10, where 10 indicates optimal performance or satisfaction. A minimal clinically significant difference is a 2-point change on the COPM performance ratings (Law et al., 2017).
Performance Quality Rating Scale - PQRS (Miller et al., 2001) | Change from baseline performance quality at 6 months
  is an observational measure of performance quality of client-selected, personally meaningful activities (therapeutic goals) originally developed for children with NDD's. The PQRS complements the COPM by assessing actual rather than perceived performances of the activities that were identified. The therapist will score each activity, using a 10-point performance rating scale between 1 (unable to perform) and 10 (performs well). The instrument is commonly used in studies involving intervention according to the CO-OP approach (Polatajko, 2017)
The Child and Adolescent Scale of Participation (CASP; Bedell, 2004). | Change from baseline participation at 6 months
  The CASP assesses children's extent of participation and restrictions in home, school and community life situations and activities compared to same-age peers as reported by family caregivers. The CASP consist of 20 items divided into four sub-sections: (1) Home participation; (2) School participation; (3) Community participation; and (4) Home and community living activities. Each item addresses a broad participation domain with examples provided for each domain. The items are rated on a 4-point scale (4 = 'Age expected/full participation', 3 = 'Somewhat limited', 2 = 'Very limited',1 = 'Unable') or as "Not applicable". There are additional open-ended questions that identify additional supports and barriers to participation. Total scores range from 0-100, with higher scores indicating better participation. The CASP was found to be f reliable and valid, with high internal consistency (α = 0.96).
Pediatric Quality of Life Inventory (PedsQL; Varni & Limbers, 2009). | Change from baseline quality of life at 6 months
  The PedsQL is used to assess health-related quality of life in children and adolescents (ages 2-18). The PedsQL consists of a 23-item in 4 domains: physical, emotional, social and school functioning. The items are rated on a 5-point scale (0 = 'Never'; 4 = 'Almost always') and linearly transformed to 0-100 scale, with higher scores indicating better health-related quality of life. The PedsQL was found to be a reliable and valid measure (high internal consistency, discriminates between groups such as children with and without a chronic condition, and responsive to change over time).

SECONDARY OUTCOMES:
Socio-Demographic and Clinical Characteristics | 1 year (before the intervention)
  Demographic and medical details will be collected from the patients' personal medical records.
Feasibility Therapist Log Book | 1-2 years (during the intervention)
  the occupational therapists who will conduct the intervention will write field notes following each session regarding the number, durations of the meetings performed, the number and reasons for cancellations cancelations. As well as the use of the key elements of the approach to ensure the implementation of the critical components of CO-OP, as described in the fidelity checklists (McEwen et al., 2012)
Parents as Partners in Intervention- Satisfaction Questionnaire - PAPI- Q (Hirsch, Waldman-Levy and Parush, 2005) | 2 years (after the intervention)
  a structured questionnaire developed in Israel designed to assess (a) parental satisfaction and involvement with occupational therapy service, for example involvement in treatment procedure, sessions attendance and general satisfaction. In the present study will ask the parents to fulfill the questionnaire following the intervention. And (b) occupational therapist following the intervention aiming to assess the levels of cooperation and involvement of the child and his family throughout the treatment process. such as their presence, participation and implementation of the guidance provided. The questioners include 17 items rank on a 1-5 Likert scale, with a higher score indicating a higher level of satisfaction. Cronbach's alpha was good (α = 0.80), suggesting that the items were inter-related and related to the scale as a whole.
Qualitative feedback interview | 2 years (after the intervention)
  a short structured interview will be conducted post intervention to obtain the parents' perception of the teleCO-OP intervention program. In the feedback interview, the parents will be asked three open-ended questions regarding a) their experience with the teleCO-OP intervention in general, b) the benefits or advantages, and c) disadvantages or barriers of this treatment method.

CONTACTS AND LOCATIONS:
Overall Officials: Yafit Gilboa, PhD, Study Director — Hebrew University of Jerusalem

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: study protocol - 1 year SAP, ICF, CSR - 3-3.5 years the data will be available until the end of the research
Access Criteria: anonyms PDF's or outputs of the statistical analysis by SPSS. the information will be sent by personal requests consider the purpose and relevant to the current research.